CLINICAL TRIAL: NCT00544557
Title: Observational Study Of The Use Of Enbrel (Registered) (Etanercept) In Routine Clinical Practice To Treat Ankylosing Spondylitis (as) Patients: An Effectiveness, Safety, And Health Economic Evaluation
Brief Title: Study Evaluating The Use Of Etanercept In Patients With Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881X1-4463; B1801087 (Other: Alias Study Number)
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Ankylosing Spondylitis
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — The patients will be treated in accordance with the requirements of the labeling of etanercept in Germany. The dosage and duration of therapy is to be determined by the physician to meet the patients' individual needs for treatment.
  Other Names: Enbrel

SUMMARY:
This study aims to provide a holistic assessment of patients receiving etanercept in a real-world setting.

DETAILED DESCRIPTION:
Non-interventional study: subjects to be selected according to the usual clinical practice of their physician

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ankylosing spondylitis (AS)

Exclusion Criteria:

* Hypersensitivity to etanercept
* Active infection including chronic or localised infection
* Sepsis or risk of sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an established diagnosis of Ankylosing Spondylitis
Sampling Method: Non-Probability Sample
Enrollment: 1715 (Actual)
Dates: Start 2007-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Klinikum Benjamin Franklin, Berlin, Germany

REFERENCES:
- [Derived] Druce KL, Aikman L, Dilleen M, Burden A, Szczypa P, Basu N. Fatigue independently predicts different work disability dimensions in etanercept-treated rheumatoid arthritis and ankylosing spondylitis patients. Arthritis Res Ther. 2018 May 29;20(1):96. doi: 10.1186/s13075-018-1598-8. PMID 29843776
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881X1-4463&StudyName=Study%20Evaluating%20The%20Use%20Of%20Etanercept%20In%20Patients%20With%20Ankylosing%20Spondylitis

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1715 participants were enrolled for documentation. Of these 1715 participants enrolled, only 1685 participants were included in analysis.
Groups:
- Etanercept: Participants who had confirmed diagnosis of ankylosing spondylitis (AS) and commenced treatment with etanercept (Enbrel) for the first time as per Summary of Product Characteristics (SmPC) were observed prospectively for 52 weeks. According to SmPC, recommended dose included etanercept 25 milligram (mg) twice weekly or 50 mg once weekly.
Period: Overall Study
Arm/Group | Etanercept
Started | 1685
Completed | 1251
Not Completed | 434
Not completed — Adverse Event | 140
Not completed — Lack of Efficacy | 196
Not completed — Other | 98

BASELINE CHARACTERISTICS:
Population: Safety population included all treated participants with available post-baseline safety data.
Arm/Group | Etanercept
Number analyzed (Participants) | 1685
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (12.9)
Sex/Gender, Customized [Number; unit: participants]
  Male | 1067
  Female | 615
  Missing | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Partial Remission at Week 26
Description: Percentage of participants achieving partial remission was determined by assessment of spondyloarthritis international society (ASAS) criteria. Partial remission was defined as a score of less than 2 units (on a scale of 0-10, where 0= no disease activity and 10= high disease activity) in each of the 4 assessment in ASAS domains: participant global assessment of disease activity, pain, function, and inflammation.
Time Frame: Week 26
Population: Effectiveness population: all treated participants greater than or equal to (>=) 18 years of age, with confirmed diagnosis of ankylosing spondylitis, who received etanercept therapy for the first time and had post-baseline documentation. Here 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1305
percentage of participants | 19.0 [16.9 to 21.2]

2. Primary Outcome: Percentage of Participants Achieving Partial Remission at Week 52
Description: Percentage of participants achieving partial remission was determined by ASAS criteria. Partial remission defined as a score of less than 2 units (on a scale of 0-10, where 0= no disease activity and 10= high disease activity) in each of the 4 assessment in ASAS domains: participant global assessment of disease activity, pain, function, and inflammation.
Time Frame: Week 52
Population: Effectiveness population: all treated participants >=18 years of age, with confirmed diagnosis of ankylosing spondylitis, who received etanercept therapy for the first time and had post-baseline documentation. Here 'N' signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1111
percentage of participants | 23.0 [20.6 to 25.6]

3. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) or Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life- threatening experience (immediate risk of dying); persistent or significant disability or incapacity; congenital anomaly. Percentage of participants with AEs included participants affected with both SAEs and non--SAEs.
Time Frame: Baseline up to Week 52
Population: Safety population included all treated participants with available post-baseline safety data.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1685
percentage of participants
  SAEs | 7.6 [20.6 to 25.6]
  AEs | 38.2

4. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) or Adverse Events (AEs) by Co-morbidity
Time Frame: Baseline up to Week 52
Population: Safety population included all treated participants with available post--baseline safety data.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1685
percentage of participants
  SAEs | NA [20.6 to 25.6] — Data was not analyzed due to low number of participants.
  AEs | NA — Data was not analyzed due to low number of participants.

5. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 52
Description: BASDAI is a validated self-assessment tool used to determine disease activity in participant with AS. Utilizing a 11-point Likert-scale (0= none and 10=very severe) participant's answered 6 questions measuring discomfort, pain and fatigue. The index was computed by adding questions 1 to 4 plus the mean of questions 5 and 6. The resulting 0 to 50 score was divided by 5 to give a final 0-10 BASDAI score (0 being no problem and 10 being the worst problem).
Time Frame: Baseline, Week 52
Population: Effectiveness population: all treated participants >=18 years of age, with confirmed diagnosis of ankylosing spondylitis, received etanercept therapy for first time and had post-baseline documentation. Here 'n' signifies participants evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
units on a scale
  Baseline (n=1635) | 5.327 (2.029)
  Change at Week 52 (n=1128) | -2.199 (2.163)

6. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 52
Description: BASFI is a validated self assessment tool that determines the degree of functional limitation in AS. Participants answered 10 questions, consisting of 8 specific questions regarding function in AS and 2 questions reflecting the participant's ability to cope with everyday life. Each question was answered on a 0-10 scale (0 being no problem and 10 being the worst problem), the sum of which (divided by 10) resulted in the BASFI score (0-10).
Time Frame: Baseline, Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
units on a scale
  Baseline (n=1626) | 4.9 (2.4)
  Change at Week 52 (n=1129) | -1.7 (2.2)

7. Secondary Outcome: Change From Baseline in Occiput-to-Wall Distance at Week 52
Description: Occiput-to-wall distance is the distance between the occiput (posterior or back portion of the head) and the wall when the participant stood with heels and shoulder against the wall and the back straight.
Time Frame: Baseline, Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
centimeter (cm)
  Baseline (n=1347) | 6.7 (7.8)
  Change at Week 52 (n=788) | -0.7 (4.4)

8. Secondary Outcome: Change From Baseline in Lateral Lumbar Flexion at Week 52
Description: Lateral lumbar flexion was determined by the difference of the finger-floor-distance in normal position and in lateral bending position.
Time Frame: Baseline, Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
cm
  Baseline (n=1123) | 11.8 (11.8)
  Change at Week 52 (n=656) | 1.0 (8.9)

9. Secondary Outcome: Change From Baseline in Patient's Global Assessment (PtGA) of Pain at Week 52
Description: Participants were asked to assess their global pain intensity within the past 7 days. Pain was evaluated on an 11-point Likert scale: min = 0 (best), max = 10 (worst).
Time Frame: Baseline, Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
units on a scale
  Baseline (n=1630) | 6.5 (2.2)
  Change at Week 52 (n=1117) | -3.0 (2.8)

10. Secondary Outcome: Change From Baseline in Patient Global Assessment (PtGA) of Disease Activity at Week 52
Description: Participants were asked to assess their disease activity within the past 7 days. Disease activity was evaluated on an 11-point Likert scale: min = 0 (best), max = 10 (worst).
Time Frame: Baseline, Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
units on a scale
  Baseline (n=1602) | 6.2 (2.3)
  Change at Week 52 (n=1094) | -3.1 (2.8)

11. Secondary Outcome: Change From Baseline in Physician Global Assessment (PGA) of Disease Activity at Week 52
Description: Physicians were asked to assess the disease activity of participants within the past 7 days. Disease activity was evaluated on an 11-point Likert scale: min = 0 (best), max = 10 (worst).
Time Frame: Baseline, Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
units on a scale
  Baseline (n=1655) | 6.4 (1.6)
  Change at Week 52 (n=1171) | -4.2 (2.2)

12. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness at Week 52
Description: Duration of morning stiffness is defined as the time elapsed when participant woke up in the morning and was able to resume normal activities without stiffness in minutes.
Time Frame: Baseline, Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
minutes
  Baseline (n=1641) | 58.6 (59.2)
  Change at Week 52 (n=1165) | -37.0 (54.0)

13. Secondary Outcome: Percentage of Participants With Significant Reduction of Morning Stiffness
Description: Duration of morning stiffness is defined as the time elapsed when participant woke up in the morning and was able to resume normal activities without stiffness in minutes. A significant reduction of duration of morning stiffness is defined as a reduction of the duration in minutes by at least 20 percent or reduction to 'no morning stiffness' (absence of morning stiffness).
Time Frame: Week 2, 6, 12, 26, 38, 52
Population: Effectiveness population: all treated participants >=18 years of age, with confirmed diagnosis of ankylosing spondylitis, received etanercept therapy for first time and had post-baseline documentation. Here 'N' signifies participants evaluable for this outcome measure and 'n' signifies participants evaluable for this measure at given time points.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
percentage of participants
  Week 2 (n=1405) | 51.6 (59.2)
  Week 6 (n=1452) | 62.1 (31.4)
  Week 12 (n=1480) | 67.2
  Week 26 (n=1395) | 68.0
  Week 38 (n=1235) | 69.8
  Week 52 (n=1186) | 70.6

14. Secondary Outcome: Percentage of Participants With Presence of Peripheral Arthritis
Description: Peripheral arthritis is the inflammation of joints that involved asymmetrically. It involved the hips, shoulder girdle (glenohumeral, acromioclavicular, and sternoclavicular joints), joints of the chest wall (costovertebral joints, costosternal junctions) and symphysis pubis.
Time Frame: Baseline, Week 2, 6, 12, 26, 38, 52
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
percentage of participants
  Baseline (n=1663) | 36.8 (59.2)
  Week 2 (n=1405) | 26.0 (31.4)
  Week 6 (n=1452) | 22.0
  Week 12 (n=1480) | 18.2
  Week 26 (n=1395) | 16.7
  Week 38 (n=1235) | 14.6
  Week 52 (n=1186) | 15.5

15. Secondary Outcome: Change From Baseline in Number of Affected Joints by Peripheral Arthritis at Week 52
Description: Peripheral arthritis is the inflammation of joints that involved asymmetrically. It involved the hips, shoulder girdle (glenohumeral, acromioclavicular, and sternoclavicular joints), joints of the chest wall (costovertebral joints, costosternal junctions) and symphysis pubis. In case of no presence of peripheral arthritis the number of affected joints was set to 0.
Time Frame: Baseline, Week 52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
joints
  Baseline (n=1652) | 2.2 (5.5)
  Change at Week 52 (n=1174) | -1.3 (5.2)

16. Secondary Outcome: Percentage of Participants With Presence of Enthesitis
Description: Enthesitis is the inflammation of the enthesis, where the joint capsules, ligaments or tendons attach to the bone. This inflammation can lead to severe pain and discomfort.
Time Frame: Baseline, Week 2, 6, 12, 26, 38, 52
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
percentage of participants
  Baseline (n=1663) | 20.6 (59.2)
  Week 2 (n=1405) | 14.7 (31.4)
  Week 6 (n=1452) | 11.5
  Week 12 (n=1480) | 9.5
  Week 26 (n=1395) | 8.5
  Week 38 (n=1235) | 7.4
  Week 52 (n=1186) | 7.9

17. Secondary Outcome: Change From Baseline in Number of Affected Body Parts by Enthesitis at Week 52
Description: Enthesitis is the inflammation of the enthesis, where the joint capsules, ligaments or tendons attach to the bone. This inflammation can lead to severe pain and discomfort. In case of no presence of enthesitis the number of affected body parts was set to 0.
Time Frame: Baseline, Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: body parts
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
body parts
  Baseline (n=1658) | 0.6 (1.6)
  Change at Week 52 (n=1174) | -0.4 (1.4)

18. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) at Week 52
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
milligram per deciliter (mg/dL)
  Baseline (n=1497) | 2.6 (4.7)
  Change at Week 52 (n=873) | -1.6 (4.4)

19. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Week 52
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 millimeter/hour (mm/hr). A higher rate is consistent with inflammation.
Time Frame: Baseline, Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
mm/hr
  Baseline (n=1422) | 26.9 (21.7)
  Change at Week 52 (n=812) | -14.2 (21.1)

20. Secondary Outcome: Percentage of Participants With Assessment in Ankylosing Spondylitis 20 (ASAS-20) Response
Description: ASAS measures symptomatic improvement in AS participants. ASAS = 4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 20= at least >= 20 percent improvement from baseline and an absolute change >=1 unit on a 0-10 numeric scale (0=no disease activity; 10=high disease activity) in at least 3 of the domains (on a 0-10 numerical scale): Global assessment of disease activity by participant, participant's global pain intensity, function measured by BASFI and inflammation measured by the average of the last two Likert-scales in BASDAI concerning morning stiffness intensity and duration and no worsening in the remaining domain.
Time Frame: Week 12, 26, 38, 52
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
percentage of participants
  Week 12 (n=1480) | 60.6 [58.0 to 63.3]
  Week 26 (n=1395) | 61.6 [58.9 to 64.3]
  Week 38 (n=1235) | 63.1 [60.3 to 66.0]
  Week 52 (n=1186) | 63.7 [60.7 to 66.5]

21. Secondary Outcome: Percentage of Participants With Assessment in Ankylosing Spondylitis 40 (ASAS-40) Response
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) participants. ASAS =4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 40= at least (>=) 40 percent improvement from baseline and an absolute change >=2 unit on a 0-10 numeric scale (0=no disease activity; 10=high disease activity) in at least 3 of the domains (on a 0-10 numerical scale): Global assessment of disease activity by participant, participant's global pain intensity, function measured by BASFI and inflammation measured by the average of the last two Likert-scales in BASDAI concerning morning stiffness intensity and duration and no worsening in the remaining domain.
Time Frame: Week 12, 26, 38, 52
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
percentage of participants
  Week 12 (n=1480) | 44.1 [41.4 to 46.8]
  Week 26 (n=1395) | 46.7 [43.9 to 49.5]
  Week 38 (n=1235) | 48.6 [45.6 to 51.5]
  Week 52 (n=1186) | 51.0 [47.9 to 54.0]

22. Secondary Outcome: Euro Quality of Life-5 Dimensions (EQ-5D) Time Trade Off (TTO)
Description: EQ 5D: participant rated questionnaire to assess health-related quality of life. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (extreme problems). Score of each domain is transformed into a single TTO value using formula developed by Greiner et al and results in a total score range -0.205 to 0.999, higher score indicates a better health state.
Time Frame: Baseline, Week 26, 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
units on a scale
  Baseline (n=1623) | 0.58 (0.30) [41.4 to 46.8]
  Week 26 (n=1343) | 0.80 (0.22) [43.9 to 49.5]
  Week 52 (n=1143) | 0.82 (0.20) [47.9 to 54.0]

23. Secondary Outcome: Euro Quality of Life (EQ--5D)- Visual Analog Scale (VAS)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life. Health. State Profile component assesses level of current health for 5 domains: mobility, self care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicate worst health state. Score of each domain is transformed into a single VAS score using formula developed by Greiner et al and results in a total score range of 0 to 100, where higher score indicates a better health state.
Time Frame: Baseline, Week 26, 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
units on a scale
  Baseline (n=1623) | 54.3 (20.7) [41.4 to 46.8]
  Week 26 (n=1343) | 71.9 (19.2) [43.9 to 49.5]
  Week 52 (n=1143) | 74.2 (18.9) [47.9 to 54.0]

24. Secondary Outcome: Work Productivity and Activity Impairment - Special Health Problems (WPAI:SHP)
Description: WPAI:SHP is 6-question participant rated questionnaire to determine the amount of absenteeism, presenteeism, work productivity loss and daily activity impairment attributable to rheumatoid arthritis for a period of 7 days prior to each visit. It yields 4 sub-scores: work time missed (absenteeism), impairment while working (presenteeism or reduced on-the-job effectiveness), overall work impairment (work productivity loss or absenteeism plus presenteeism) and activity impairment (daily activity impairment). These sub-scores are transformed to impairment percentages (range from 0 to 100), with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline, Week 26, 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
percentage of impairment
  Baseline: Work Time Missed (n=776) | 21.9 (36.3) [41.4 to 46.8]
  Baseline: Impairment While Working (n=890) | 48.3 (26.9) [43.9 to 49.5]
  Baseline: Overall work impairment (n=716) | 52.9 (29.8) [47.9 to 54.0]
  Baseline: Activity impairment (n = 1624) | 58.1 (24.6)
  Week 26: Work Time Missed (n = 666) | 6.6 (20.6)
  Week 26: Impairment While Working (n = 799) | 27.3 (23.1)
  Week 26: Overall work impairment (n = 657) | 29.8 (25.9)
  Week 26: Activity impairment (n = 1331) | 34.6 (24.6)
  Week 52: Work Time Missed (n = 588) | 6.3 (19.2)
  Week 52: Impairment While Working (n = 706) | 24.6 (21.9)
  Week 52: Overall work impairment (n = 578) | 26.3 (24.2)
  Week 52: Activity impairment (n = 1137) | 32.3 (24.9)

25. Secondary Outcome: Healthcare Resource Utilization
Description: Participants utilization of healthcare resources was evaluated as number of events for healthcare resources utilization including: number of visits to general practitioners, visits to rheumatologist, visits to other medical specialists, inpatient hospitalizations, inpatient rehabilitations, inpatient follow-up treatment, outpatient rehabilitations, physiotherapy, and other healthcare utilizations. At baseline, number of events for participants' healthcare resources utilization during last 12 months before enrollment into the study were documented. After enrollment, number of events for participants' healthcare resources utilization were documented for last 6 months after previous documentation.
Time Frame: Baseline, Week 26, 52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
events
  Baseline: General Practitioner Visit (n=1654) | 4.7 (8.3) [41.4 to 46.8]
  Baseline: Rheumatologist Visit (n=1657) | 3.7 (3.3) [43.9 to 49.5]
  Baseline: Other Specialist Visit (n=1659) | 1.6 (3.1) [47.9 to 54.0]
  Baseline: In-patient Hospitalization (n = 1658) | 0.3 (0.9)
  Baseline: In-patient Rehabilitation (n = 1657) | 0.2 (1.6)
  Baseline: Follow-up Treatment (n = 1662) | 0.0 (0.1)
  Baseline: Out-patient Rehabilitation (n = 1661) | 0.0 (0.8)
  Baseline: Physiotherapy (n = 1659) | 9.1 (25.0)
  Baseline: Out-patient Hospitalization (n = 1663) | 0.0 (0.1)
  Baseline: Ergotherapy (n = 1663) | 0.0 (0.1)
  Baseline: Other Health Care Resources (n = 1662) | 0.7 (7.4)
  Baseline: Sum Over All Care Resources (n = 1663) | 20.3 (29.7)
  Week 26: General Practitioner Visit (n = 1389) | 2.2 (3.1)
  Week 26: Rheumatologist Visit (n = 1392) | 3.0 (2.6)
  Week 26: Other Specialist Visit (n = 1393) | 0.6 (1.5)
  Week 26: In-patient Hospitalization (n = 1395) | 0.1 (0.6)
  Week 26: In-patient Rehabilitation (n = 1392) | 0.2 (1.9)
  Week 26: Follow-up Treatment (n = 1395) | 0.0 (0.2)
  Week 26: Out-patient Rehabilitation (n = 1395) | 0.0 (0.8)
  Week 26: Physiotherapy (n = 1395) | 5.0 (14.1)
  Week 26: Out-patient Hospitalization (n = 1394) | 0.0 (0.0)
  Week 26: Ergotherapy (n = 1395) | 0.0 (0.5)
  Week 26: Other Health Care Resources (n = 1390) | 0.5 (4.5)
  Week 26: Sum Over All Care Resources (n = 1395) | 11.5 (16.9)
  Week 52: General Practitioner Visit (n = 1184) | 1.8 (3.8)
  Week 52: Rheumatologist Visit (n = 1184) | 2.0 (1.9)
  Week 52: Other Specialist Visit (n = 1183) | 0.6 (2.6)
  Week 52: In-patient Hospitalization (n = 1186) | 0.0 (0.2)
  Week 52: In-patient Rehabilitation (n = 1186) | 0.1 (0.9)
  Week 52: Follow-up Treatment (n = 1186) | 0.0 (0.0)
  Week 52: Out-patient Rehabilitation (n = 1186) | 0.0 (0.7)
  Week 52: Physiotherapy (n = 1186) | 4.3 (13.3)
  Week 52: Out-patient Hospitalization (n = 1186) | 0.0 (0.0)
  Week 52: Ergotherapy (n = 1186) | 0.0 (0.9)
  Week 52: Other Health Care Resources (n = 1185) | 0.7 (5.1)
  Week 52: Sum Over All Care Resources (n = 1186) | 9.6 (15.8)

26. Secondary Outcome: Duration of Healthcare Resources Utilization
Description: Participants duration of healthcare resources utilization was evaluated as number of days for healthcare resources utilization including: duration of visits to general practitioners, to rheumatologist, to other medical specialists, inpatient hospitalizations, inpatient rehabilitations, inpatient follow-up treatment, outpatient rehabilitations, physiotherapy, and other healthcare utilizations. At baseline, number of days for participants' healthcare resources utilizations during last 12 months before enrollment into the study were documented. After enrollment, number of days for participants' healthcare resources utilization were documented for last 6 months after previous documentation.
Time Frame: Baseline, Week 26, 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Etanercept
Number analyzed (Participants) | 1663
days
  Baseline: General Practitioner Visit (n=986) | 3.7 (10.5) [41.4 to 46.8]
  Baseline: Rheumatologist Visit (n=928) | 3.1 (5.7) [43.9 to 49.5]
  Baseline: Other Specialist Visit (n=1242) | 0.9 (2.5) [47.9 to 54.0]
  Baseline: In-patient Hospitalization (n = 1633) | 2.0 (5.7)
  Baseline: In-patient Rehabilitation (n = 1648) | 1.5 (6.0)
  Baseline: Follow-up Treatment (n = 1661) | 0.1 (1.8)
  Baseline: Out-patient Rehabilitation (n = 1654) | 0.2 (3.6)
  Baseline: Physiotherapy (n = 1551) | 6.2 (20.2)
  Baseline: Out-patient Hospitalization (n = 1661) | 0.0 (0.0)
  Baseline: Ergotherapy (n = 1663) | 0.0 (0.1)
  Baseline: Other Health Care Resources (n = 1641) | 0.4 (6.0)
  Baseline: Sum Over All Care Resources (n = 1663) | 14.5 (28.0)
  Week 26: General Practitioner Visit (n = 917) | 1.2 (2.1)
  Week 26: Rheumatologist Visit (n = 834) | 2.2 (2.7)
  Week 26: Other Specialist Visit (n = 1190) | 0.4 (1.9)
  Week 26: In-patient Hospitalization (n = 1390) | 0.3 (1.9)
  Week 26: In-patient Rehabilitation (n = 1391) | 1.0 (5.1)
  Week 26: Follow-up Treatment (n = 1395) | 0.0 (0.6)
  Week 26: Out-patient Rehabilitation (n = 1394) | 0.1 (1.2)
  Week 26: Physiotherapy (n = 1350) | 3.0 (9.9)
  Week 26: Out-patient Hospitalization (n = 1395) | 0.0 (0.0)
  Week 26: Ergotherapy (n = 1393) | 0.0 (0.4)
  Week 26: Other Health Care Resources (n = 1376) | 0.3 (4.0)
  Week 26: Sum Over All Care Resources (n = 1395) | 7.0 (14.5)
  Week 52: General Practitioner Visit (n = 762) | 1.0 (1.7)
  Week 52: Rheumatologist Visit (n = 716) | 1.5 (2.1)
  Week 52: Other Specialist Visit (n = 1009) | 0.3 (2.3)
  Week 52: In-patient Hospitalization (n = 1177) | 0.3 (2.0)
  Week 52: In-patient Rehabilitation (n = 1185) | 0.4 (3.0)
  Week 52: Follow-up Treatment (n = 1186) | 0.0 (0.0)
  Week 52: Out-patient Rehabilitation (n = 1186) | 0.2 (3.7)
  Week 52: Physiotherapy (n = 1151) | 2.6 (9.6)
  Week 52: Out-patient Hospitalization (n = 1186) | 0.0 (0.0)
  Week 52: Ergotherapy (n = 1186) | 0.0 (0.9)
  Week 52: Other Health Care Resources (n = 1162) | 0.2 (2.5)
  Week 52: Sum Over All Care Resources (n = 1186) | 5.4 (13.9)

27. Secondary Outcome: Percentage of Participants With Prior or Concomitant Medication Use for Treatment of Ankylosing Spondylitis
Description: Participants taking any non-study medications which were administered either prior to or during the study treatment for AS were reported.
Time Frame: Baseline up to Week 52
Population: Safety population included all treated participants with available post-baseline safety data.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1685
percentage of participants
  Concomitant Medication | 38.4 [58.0 to 63.3]
  Prior Therapy | 98.6 [60.7 to 66.5]

28. Secondary Outcome: Percentage of Participants With Discontinuation of Treatment Due to Adverse Events
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Baseline up to Week 52
Population: Safety population included all treated participants with available post--baseline safety data.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1685
percentage of participants | 11.8

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as non-serious in another subject, or one subject may have experienced both a serious and non-serious event during the study.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 128/1685
Other Adverse Events (participants affected / at risk) | 588/1685
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=1685)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 7
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2
Spondylitis (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intracranial haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oropharyngeal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pneumonia (Infections and infestations) | 3
Abdominal abscess (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Campylobacter gastroenteritis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Meningitis aseptic (Infections and infestations) | 1
Meningitis viral (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 2
Joint dislocation (Injury, poisoning and procedural complications) | 2
Tendon rupture (Injury, poisoning and procedural complications) | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1
Lymphatic duct rupture (Injury, poisoning and procedural complications) | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Sports injury (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Crohn's disease (Gastrointestinal disorders) | 4
Inguinal hernia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1
Papilla of Vater stenosis (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Migraine with aura (Nervous system disorders) | 2
Aphasia (Nervous system disorders) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Demyelination (Nervous system disorders) | 1
Dysaesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Hemianopia homonymous (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Monoplegia (Nervous system disorders) | 1
Movement disorder (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Thalamic infarction (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Coronary artery disease (Cardiac disorders) | 4
Myocardial infarction (Cardiac disorders) | 4
Angina pectoris (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Condition aggravated (General disorders) | 5
Drug ineffective (General disorders) | 2
Oedema peripheral (General disorders) | 2
Pain (General disorders) | 2
Impaired healing (General disorders) | 1
Injection site hypersensitivity (General disorders) | 1
Hip surgery (Surgical and medical procedures) | 1
Implantable defibrillator insertion (Surgical and medical procedures) | 1
Inguinal hernia repair (Surgical and medical procedures) | 1
Myringoplasty (Surgical and medical procedures) | 1
Removal of foreign body (Surgical and medical procedures) | 1
Spinal fusion surgery (Surgical and medical procedures) | 1
Tonsillectomy (Surgical and medical procedures) | 1
Cholangitis (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 2
Bile duct stone (Hepatobiliary disorders) | 1
Biliary colic (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Psychogenic pain disorder (Psychiatric disorders) | 2
Acute stress disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 2
Renal colic (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 2
Haematoma (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Iritis (Eye disorders) | 2
Cataract (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Maculopathy (Eye disorders) | 1
Goitre (Endocrine disorders) | 3
Arthroscopy (Investigations) | 1
Transaminases increased (Investigations) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Bone marrow disorder (Blood and lymphatic system disorders) | 1
Skull malformation (Congenital, familial and genetic disorders) | 1
Sarcoidosis (Immune system disorders) | 1
Cervical polyp (Reproductive system and breast disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=1685)
Nasopharyngitis (Infections and infestations) | 59
Bronchitis (Infections and infestations) | 32
Upper respiratory tract infection (Infections and infestations) | 24
Infection (Infections and infestations) | 13
Sinusitis (Infections and infestations) | 9
Urinary tract infection (Infections and infestations) | 9
Oral herpes (Infections and infestations) | 8
Respiratory tract infection (Infections and infestations) | 8
Pharyngitis (Infections and infestations) | 7
Febrile infection (Infections and infestations) | 6
Cystitis (Infections and infestations) | 5
Herpes simplex (Infections and infestations) | 5
Herpes zoster (Infections and infestations) | 5
Bronchopneumonia (Infections and infestations) | 4
Ear infection (Infections and infestations) | 4
Furuncle (Infections and infestations) | 4
Otitis media (Infections and infestations) | 4
Rhinitis (Infections and infestations) | 4
Tonsillitis (Infections and infestations) | 4
Acute tonsillitis (Infections and infestations) | 3
Laryngitis (Infections and infestations) | 3
Erysipelas (Infections and infestations) | 2
Folliculitis (Infections and infestations) | 2
Fungal skin infection (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Genital herpes (Infections and infestations) | 1
Infection susceptibility increased (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Rash pustular (Infections and infestations) | 2
Streptococcal infection (Infections and infestations) | 2
Tracheobronchitis (Infections and infestations) | 2
Acarodermatitis (Infections and infestations) | 1
Cellulitis of male external genital organ (Infections and infestations) | 1
Erythrasma (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Gastrointestinal candidiasis (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Genital candidiasis (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Injection site infection (Infections and infestations) | 1
Oophoritis (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pseudofolliculitis barbae (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Vaginal candidiasis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Viral tonsillitis (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Wound infection staphylococcal (Infections and infestations) | 1
Injection site erythema (General disorders) | 69
Injection site pruritus (General disorders) | 21
Injection site reaction (General disorders) | 25
Condition aggravated (General disorders) | 20
Fatigue (General disorders) | 14
Injection site swelling (General disorders) | 13
Injection site irritation (General disorders) | 10
Oedema peripheral (General disorders) | 9
Pyrexia (General disorders) | 9
Injection site hypersensitivity (General disorders) | 5
Chest pain (General disorders) | 4
Local swelling (General disorders) | 4
Drug ineffective (General disorders) | 3
Drug intolerance (General disorders) | 3
General physical health deterioration (General disorders) | 3
Impaired healing (General disorders) | 3
Injection site pain (General disorders) | 3
Injection site urticaria (General disorders) | 3
Pain (General disorders) | 3
Injection site induration (General disorders) | 2
Injection site macule (General disorders) | 2
Injection site warmth (General disorders) | 2
Tenderness (General disorders) | 2
Application site erythema (General disorders) | 1
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 1
Feeling hot (General disorders) | 1
Granuloma (General disorders) | 1
Injection site dermatitis (General disorders) | 1
Injection site discolouration (General disorders) | 1
Injection site necrosis (General disorders) | 1
Injection site oedema (General disorders) | 1
Injection site paraesthesia (General disorders) | 1
Injection site rash (General disorders) | 1
Local reaction (General disorders) | 1
Localised oedema (General disorders) | 1
Malaise (General disorders) | 1
Sensation of foreign body (General disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 18
Acne (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3
Blister (Skin and subcutaneous tissue disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 9
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 8
Erythema (Skin and subcutaneous tissue disorders) | 17
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1
Generalised erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Nail psoriasis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 10
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 10
Rash generalised (Skin and subcutaneous tissue disorders) | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 3
Skin reaction (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 2
Petechiae (Skin and subcutaneous tissue disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin induration (Skin and subcutaneous tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1
Skin nodule (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 16
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7
Joint swelling (Musculoskeletal and connective tissue disorders) | 6
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Enthesopathy (Musculoskeletal and connective tissue disorders) | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myosclerosis (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3
Tendonitis (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Joint effusion (Musculoskeletal and connective tissue disorders) | 2
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 1
Dactylitis (Musculoskeletal and connective tissue disorders) | 1
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Gouty tophus (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 19
Nausea (Gastrointestinal disorders) | 19
Abdominal pain (Gastrointestinal disorders) | 7
Crohn's disease (Gastrointestinal disorders) | 4
Colitis ulcerative (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 3
Periodontitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 2
Gingival pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Anal fissure (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Breath odour (Gastrointestinal disorders) | 1
Chapped lips (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Epiploic appendagitis (Gastrointestinal disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Lip dry (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Radicular cyst (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Stomach discomfort (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 18
Dizziness (Nervous system disorders) | 11
Paraesthesia (Nervous system disorders) | 5
Carpal tunnel syndrome (Nervous system disorders) | 4
Sciatica (Nervous system disorders) | 4
Syncope (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 3
Cervical root pain (Nervous system disorders) | 2
Cervicobrachial syndrome (Nervous system disorders) | 2
Movement disorder (Nervous system disorders) | 2
Sensory disturbance (Nervous system disorders) | 2
Amnesia (Nervous system disorders) | 1
Areflexia (Nervous system disorders) | 1
Autonomic nervous system imbalance (Nervous system disorders) | 1
Dysaesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Hyperaesthesia (Nervous system disorders) | 1
Intercostal neuralgia (Nervous system disorders) | 1
Meralgia paraesthetica (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope vasovagal (Nervous system disorders) | 1
Alanine aminotransferase increased (Investigations) | 9
Gamma-glutamyltransferase increased (Investigations) | 7
Liver function test abnormal (Investigations) | 6
Hepatic enzyme increased (Investigations) | 4
Blood alkaline phosphatase increased (Investigations) | 3
Haemoglobin decreased (Investigations) | 3
Transaminases increased (Investigations) | 3
Weight increased (Investigations) | 3
Arthroscopy (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Investigation (Investigations) | 2
Antinuclear antibody positive (Investigations) | 1
Bacterial test positive (Investigations) | 1
Biopsy prostate (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood urine present (Investigations) | 1
C-reactive protein increased (Investigations) | 1
DNA antibody positive (Investigations) | 1
Diagnostic procedure (Investigations) | 1
ECG signs of myocardial ischaemia (Investigations) | 1
Heart rate increased (Investigations) | 1
Laboratory test abnormal (Investigations) | 1
Lipase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Red blood cell sedimentation rate increased (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Blood pressure diastolic increased (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1
Iritis (Eye disorders) | 9
Visual disturbance (Eye disorders) | 4
Conjunctivitis (Eye disorders) | 3
Ocular hyperaemia (Eye disorders) | 3
Uveitis (Eye disorders) | 3
Abnormal sensation in eye (Eye disorders) | 2
Cataract (Eye disorders) | 2
Dry eye (Eye disorders) | 2
Iridocyclitis (Eye disorders) | 2
Diplopia (Eye disorders) | 1
Eye swelling (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Hospitalisation (Surgical and medical procedures) | 4
Carpal tunnel decompression (Surgical and medical procedures) | 2
Synoviorthesis (Surgical and medical procedures) | 2
Abortion induced (Surgical and medical procedures) | 1
Angioplasty (Surgical and medical procedures) | 1
Ankle operation (Surgical and medical procedures) | 1
Arterial stent insertion (Surgical and medical procedures) | 1
Baker's cyst excision (Surgical and medical procedures) | 1
Cataract operation (Surgical and medical procedures) | 1
Catheterisation cardiac (Surgical and medical procedures) | 1
Dental operation (Surgical and medical procedures) | 1
Dental treatment (Surgical and medical procedures) | 1
Hip arthroplasty (Surgical and medical procedures) | 1
Infiltration anaesthesia (Surgical and medical procedures) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Ligament operation (Surgical and medical procedures) | 1
Neurolysis (Surgical and medical procedures) | 1
Osteotomy (Surgical and medical procedures) | 1
Skin operation (Surgical and medical procedures) | 1
Spinal deformity correction (Surgical and medical procedures) | 1
Surgery (Surgical and medical procedures) | 1
Tendon operation (Surgical and medical procedures) | 1
Tendon sheath incision (Surgical and medical procedures) | 1
Tonsillectomy (Surgical and medical procedures) | 1
Tooth extraction (Surgical and medical procedures) | 1
Fall (Injury, poisoning and procedural complications) | 7
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 3
Meniscus lesion (Injury, poisoning and procedural complications) | 3
Accident (Injury, poisoning and procedural complications) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1
Skin injury (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Hypertension (Vascular disorders) | 8
Cardiovascular insufficiency (Vascular disorders) | 2
Thrombosis (Vascular disorders) | 2
Haematoma (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Varicose vein (Vascular disorders) | 1
Depression (Psychiatric disorders) | 5
Depressed mood (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Agitation (Psychiatric disorders) | 1
Alcohol abuse (Psychiatric disorders) | 1
Libido decreased (Psychiatric disorders) | 1
Mood swings (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Somatoform disorder (Psychiatric disorders) | 1
Tobacco abuse (Psychiatric disorders) | 1
Angina pectoris (Cardiac disorders) | 3
Cardiovascular disorder (Cardiac disorders) | 2
Coronary artery disease (Cardiac disorders) | 2
Mitral valve incompetence (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 2
Bradycardia (Cardiac disorders) | 1
Cardiac discomfort (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Mitral valve prolapse (Cardiac disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 6
Delivery (Pregnancy, puerperium and perinatal conditions) | 1
First trimester pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Hypersensitivity (Immune system disorders) | 4
Sarcoidosis (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Gout (Metabolism and nutrition disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Cow's milk intolerance (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Anaemia macrocytic (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Ear pruritus (Ear and labyrinth disorders) | 1
Inner ear inflammation (Ear and labyrinth disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Calculus urinary (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 3
Genital erythema (Reproductive system and breast disorders) | 1
Menstruation irregular (Reproductive system and breast disorders) | 1
Androgen deficiency (Endocrine disorders) | 1
Cushing's syndrome (Endocrine disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Campylobacter infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.